CLINICAL TRIAL: NCT01133236
Title: Randomized Clinical Trial to Assess the Effect of Fluid and Salt Restriction on the Management of Patients Hospitalized Due to Decompensated Heart Failure
Brief Title: Fluid and Salt Restriction in Decompensated Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Eneida Rejane Rabelo da Silva, Professor, PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS and HCPA 09117
Record Dates: First submitted 2009-11-09; First posted 2010-05-28 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure
Keywords: Salt restriction; Fluid restriction; Congestion; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Salts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salt and Fluid (Experimental): Intervention: Fluid 800 Ml and Salt 2 g per day Control: FLuid and Salt Free
  Interventions: Dietary Supplement: Salt and fluid restriction

INTERVENTIONS:
Dietary Supplement: Salt and fluid restriction — I: Intervention Prescription of low-sodium diet with additional 2 g of sodium and water restriction to 800 mL/day.
  II: Control Prescription without sodium and fluid restriction.

SUMMARY:
The non-pharmacological measures that are widely practiced and recommended for HF patients, such as salt and water restriction, specially at moments of disease decompensation, still lack clearer evidence of their therapeutic effect.

DETAILED DESCRIPTION:
Heart Failure Clinics, healthcare structures formed by a multidisciplinary team specialized in the disease, have demonstrated to provide benefits to patients through multiple non-pharmacological interventions, among them fluid and salt restriction. Sodium restriction has a class I recommendation and evidence level C, that is, general agreement that the intervention is beneficial, useful and effective, evidenced by consensus, expert opinion, small studies, retrospective studies or registries. Sodium restriction becomes even more controversial when we consider evidence suggesting the benefit of non-salt restriction or treatments with salt administration, in the form of hypertonic solutions. In face of literature evidence not showing conclusive results about the benefit of sodium and fluid restriction, we designed this study in order to assess the effect of fluid and salt restriction on the management of patients hospitalized due to decompensated heart failure

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, with age equal to or above 18 years, diagnosed with decompensated HR (systolic dysfunction), according to the Boston Criteria (score > 8 points), who agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Patients presenting with endogenous creatinine clearance (ECC) values lower than or equal to 50-60 mL/min (obtained by the Cockcroft-Gault equation) at hospital admission, cardiogenic shock, survival compromised by another evolving disease, those with difficulty complying with treatment (dementia, cognitive deficit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Bodyweight loss | 7 days
  Daily weight on a digital scale
Clinical stability | Seven days.
  Clinical assessment daily for 7 days.

SECONDARY OUTCOMES:
Health state evaluation. | 30 days
  Evaluation of health state using the Euro-QOL 5D for 30 days after the 7th day of clinical stability assessment.
Evaluation of thirst sensation. | Seven days
  Evaluation of thirst score on the Thirst Scale, daily for seven days.
Re-hospitalizations. | 30 days
  Medical records assessed for 30 days after the 7th day of clinical stability assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis B Silva-Neto, MD, ScD, Principal Investigator — Post Graduated Program of Federal University Program

REFERENCES:
- [Derived] Aliti GB, Rabelo ER, Clausell N, Rohde LE, Biolo A, Beck-da-Silva L. Aggressive fluid and sodium restriction in acute decompensated heart failure: a randomized clinical trial. JAMA Intern Med. 2013 Jun 24;173(12):1058-64. doi: 10.1001/jamainternmed.2013.552. PMID 23689381